CLINICAL TRIAL: NCT03845114
Title: Reduction of Basal Insulin to Prevent Hypoglycemia During Two Types of Exercise in Adults and Adolescents With Type 1 Diabetes Using Insulin Pump Therapy
Brief Title: Insulin-based Strategies to Prevent Hypoglycemia During Two Types of Exercise
Acronym: RIDE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RIDE-2
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 diabetes; Exercise; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Continuous exercise - Basal insulin reduced by 40% (Active Comparator)
  Interventions: Other: Continous exercise; Other: Reduction of basal insulin by 40%
- Continuous exercise - Basal insulin reduced by 80% (Active Comparator)
  Interventions: Other: Continous exercise; Other: Reduction of basal insulin by 80%
- Interval exercise - Basal insulin reduced by 40% (Active Comparator)
  Interventions: Other: Interval exercise; Other: Reduction of basal insulin by 40%
- Interval exercise - Basal insulin reduced by 80% (Active Comparator)
  Interventions: Other: Interval exercise; Other: Reduction of basal insulin by 80%

INTERVENTIONS:
Other: Continous exercise — 60-minute continuous exercise on the ergocycle at 60% of VO2 peak (moderate intensity).
  Arms: Continuous exercise - Basal insulin reduced by 40%; Continuous exercise - Basal insulin reduced by 80%
Other: Interval exercise — Participants will perform a 60-minute interval exercise on the ergocycle at 60% of VO2 peak (moderate intensity).
  Arms: Interval exercise - Basal insulin reduced by 40%; Interval exercise - Basal insulin reduced by 80%
Other: Reduction of basal insulin by 40% — Participant's insulin basal rate will be reduced by 40% 1 hour before exercise onset.
  Arms: Continuous exercise - Basal insulin reduced by 40%; Interval exercise - Basal insulin reduced by 40%
Other: Reduction of basal insulin by 80% — Participant's insulin basal rate will be reduced by 80% 1 hour before exercise onset.
  Arms: Continuous exercise - Basal insulin reduced by 80%; Interval exercise - Basal insulin reduced by 80%

SUMMARY:
Regular exercise is associated with many health benefits for individuals with type 1 diabetes. However, immediate and delayed exercise-induced hypoglycemia is frequent and thus the main limiting factor for physical activity practice in this population. To reduce the risk of exercise-induced hypoglycemia, two types of adjustments may be considered by patients with type 1 diabetes : pre-meal insulin-dose reduction and carbohydrate supplements. Few evidence-based recommendations are available for patients using insulin pump to adjust insulin doses in order to limit exercise-induced hypoglycemia. The objective of this study is to address the magnitude of the needed reduction during two types of frequently practiced exercise (continuous vs. interval exercise) known to have a different impact on blood glucose reduction.

DETAILED DESCRIPTION:
Each study participant will be admitted at IRCM one to five days after sensor insertion. Participants will be asked to change their pump catheter 24 to 36 hours prior to the intervention visit. On the day of the intervention visit, participants will have a standardized lunch (45-65g CHO for females and 60-80g CHO for males ) at 12:00 and will be asked not to eat afterwards (except for correction of hypoglycemia). Participants will be asked not to exercise (excluding light exercise such as walking or taking the stairs) the day before and the day of the intervention visit. Participants will be asked not to consume caffeine after 12:00 the day of the intervention. The day before the intervention and the day of the intervention, participants will be asked to refrain from alcohol consumption. Participants will be blinded to the strategy used during the exercise intervention. Participants will be admitted at IRCM at 14:00. A catheter will be installed for plasma glucose and insulin measurements. At 14:30, insulin basal rate will be reduced by 40% or 80% depending of randomization. At 15:30, participants will undertake a continuous exercise (60-minute exercise on the ergocycle at 60% of VO2 peak) or an interval exercise (2-minutes alternating intervals at 85% and 50% of VO2peak for 50-minutes, with 5-minutes at 45% VO2peak at the start and the end of exercise). As a safety measure, plasma glucose will be measured every 10 minutes. Participants will be blinded to sensor glucose levels as well as plasma glucose measurements. At 17:00, the participant will be discharged if glucose levels are above 5.5 mmol/L. Participants will be asked to eat a standardized dinner at home (45-65g CHO for females and 60-80g CHO for males). Participants will have the freedom to choose at what time they wish to have dinner but it will have to be similar on all intervention visits.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 14 years of old.
2. Clinical diagnosis of type 1 diabetes for at least two years.
3. The subject will have been on insulin pump therapy for at least 3 months.
4. Last (less than 2 months) HbA1c ≤ 10%.

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy or severe proliferative retinopathy as judged by the investigator.
2. Recent (< 3 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Abnormal blood panel and/or anemia.
4. Ongoing pregnancy.
5. Severe hypoglycemic episode within two weeks of screening.
6. Other serious medical illness likely to interfere with study participation or with the ability to complete the exercise periods by the judgment of the investigator (e.g. orthopedic limitation).
7. Failure to comply with team's recommendations (e.g. not willing to change pump parameters, etc.).

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-06-30 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Decrease in plasma glucose levels during exercise | 60 minutes
  Difference between glucose levels at the beginning of the exercise and the lowest glucose levels from the start of the exercise until the end of exercise

SECONDARY OUTCOMES:
Percentage of time of plasma glucose levels spent below 4 mmol/L | 60 minutes
Decremental area under the curve of plasma glucose levels | 60 minutes
Area under the curve of plasma glucose levels < 4 mmol/L | 60 minutes
Number of patients with an exercise-induced hypoglycemia < 3.9 mmol/L | 60 minutes
Number of patients with an exercise-induced hypoglycemia < 3.5 mmol/L | 60 minutes
Number of patients requiring an oral treatment for hypoglycemia | 60 minutes
Total number of hypoglycemia episodes requiring treatment | 60 minutes
Percentage of time of plasma glucose levels spent > 10 mmol/L | 60 minutes
Percentage of time of plasma glucose levels spent between 4-10 mmol/L | 60 minutes
Mean time to the first hypoglycemic event | 60 minutes
Amount of carbohydrates needed to treat a hypoglycemic event | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (2):
- Canada (2):
  - Institut de recherches cliniques de Montréal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec